CLINICAL TRIAL: NCT02865824
Title: Effects of Antiplatelets Discontinuation in Patients Receiving Polypectomy: Randomized Controlled Trial
Brief Title: Polypectomy in Patients Taking Dual Antiplatelet Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Joon Sung Kim, Doctor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC
Record Dates: First submitted 2016-08-01; First posted 2016-08-15 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Colonic Polyps
Keywords: Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continue thienopyridine (Active Comparator): Patients continue dual antiplatelet therapy (DAT) before colonoscopy and all polyps are removed by cold snare polypectomy.
  Interventions: Drug: Continue thienopyridine
- Discontinue thienopyridine (Experimental): Patients discontinue thienopyridines for 1 week before colonoscopy and all polyps are removed by cold snare polypectomy.
  Interventions: Drug: Discontinue thienopyridine

INTERVENTIONS:
Drug: Continue thienopyridine — Patients continue dual antiplatelet therapies before colonoscopy. The patients continue taking thienopyridine before colonoscopy
  Other Names: DAT group
  Arms: Continue thienopyridine
Drug: Discontinue thienopyridine — Patients who are taking dual antiplatelet therapies stop thienopyridine one week before they undergo colonoscopy
  Other Names: Aspirin group
  Arms: Discontinue thienopyridine

SUMMARY:
Current guidelines recommend discontinuation of antiplatelets (i.e clopidogrel) for 7 days in patients taking DAT (dual antiplatelet therapy) before colonoscopy and polypectomy. The purpose of this study was to examine if a) discontinuation of these drugs reduces bleeding risks during polypectomy and if b) discontinuation of these drugs increases the occurence of thromboembolic events.

DETAILED DESCRIPTION:
Patients taking dual antiplatelets (DAT) and who visited for colonoscopy were eligible for enrollment in this study. On enrollment, patients were randomized to two groups. One group continued DAT and the other group discontinued antiplatelets (i.e. clopidogrel, ticagrelor, prasugrel) for 7 days before colonoscopy. If polyps (≤1 cm) were observed during colonoscopy, they were removed by cold snare polypectomy. The primary aim was to compared the delayed bleeding rates of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 20 years undergoing routine colonoscopy
* patients who are taking DAT (dual antiplatelet therapy)

Exclusion Criteria:

* patients not abiding to the study protocol
* history of inflammatory bowel disease
* severe comorbidities
* American Society of Anesthesiology class III or more
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Delayed bleeding requiring hemostasis after polypectomy | 2 weeks

SECONDARY OUTCOMES:
immediate bleeding requiring hemostasis after polypectomy | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Joon Sung Kim, MD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Incheon St. Mary's Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Won D, Kim JS, Ji JS, Kim BW, Choi H. Cold Snare Polypectomy in Patients Taking Dual Antiplatelet Therapy: A Randomized Trial of Discontinuation of Thienopyridines. Clin Transl Gastroenterol. 2019 Oct;10(10):e00091. doi: 10.14309/ctg.0000000000000091. PMID 31599746